CLINICAL TRIAL: NCT00237640
Title: Effect of Cinnamon on Glucose and Lipid Levels in Non-Insulin Dependent Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11798
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Adult Onset
Keywords: Cinnamon; Diabetes mellitus; Hyperlipidemia; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperlipidemias; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Cinnamon or placebo 500 mg capsule twice daily
- 2 (Active Comparator)
  Interventions: Drug: Cinnamon or placebo 500 mg capsule twice daily

INTERVENTIONS:
Drug: Cinnamon or placebo 500 mg capsule twice daily — Cinnamon 500 mg capsule twice daily or placebo capsule twice daily

SUMMARY:
The purpose of this study is to determine the effects of cinnamon on serum glucose and lipid levels in people with non-insulin dependent type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Forty people with non-insulin dependent type 2 diabetes mellitus will be randomized to receive either cinnamon or placebo for three months. The dose of cinnamon will be one gram daily. Fasting serum glucose, triglyceride, total cholesterol, LDL, HDL, and insulin levels will be measured at baseline and at 1, 2, and 3 months. HbA1c levels will be measured at baseline and at 3 months. Patients will be monitored for compliance, adverse effects, and dietary changes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* HbA1C > 6.0%
* Age 18 and above
* Able to obtain consent

Exclusion Criteria:

* Currently taking insulin
* Pregnancy
* End-stage renal disease
* Hemolytic anemia
* Cinnamon intolerance
* Inability or unwillingness to adhere to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
- Primary outcomes include HbA1c, glucose, total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides levels. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Steve M Blevins, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- General Clinical Research Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Blevins SM, Leyva MJ, Brown J, Wright J, Scofield RH, Aston CE. Effect of cinnamon on glucose and lipid levels in non insulin-dependent type 2 diabetes. Diabetes Care. 2007 Sep;30(9):2236-7. doi: 10.2337/dc07-0098. Epub 2007 Jun 11. No abstract available. PMID 17563345